CLINICAL TRIAL: NCT01307579
Title: A Randomized Open-Label Trial of Caspofungin Versus Fluconazole to Prevent Invasive Fungal Infections in Children Undergoing Chemotherapy for Acute Myeloid Leukemia (AML)
Brief Title: Caspofungin Versus Fluconazole in Preventing Invasive Fungal Infections (IFI) in Patients Undergoing Chemotherapy for Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ACCL0933; NCI-2011-02640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000695748; COG-ACCL0933; S12-00316; ACCL0933 (Other: Childrens Oncology Group); COG-ACCL0933 (Other: DCP); ACCL0933 (Other: CTEP); U10CA095861 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2019-06

CONDITIONS: Acute Myeloid Leukemia; Adult Acute Monoblastic Leukemia; Adult Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With Maturation; Adult Acute Myeloid Leukemia With Minimal Differentiation; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22.3;q23.3); MLLT3-KMT2A; Adult Acute Myeloid Leukemia Without Maturation; Adult Acute Myelomonocytic Leukemia; Alkylating Agent-Related Acute Myeloid Leukemia; Childhood Acute Monoblastic Leukemia; Childhood Acute Monocytic Leukemia; Childhood Acute Myeloid Leukemia in Remission; Childhood Acute Myeloid Leukemia With Maturation; Childhood Acute Myeloid Leukemia With Minimal Differentiation; Childhood Acute Myeloid Leukemia Without Maturation; Childhood Acute Myelomonocytic Leukemia; Fungal Infection; Myeloid Neoplasm; Neutropenia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia; Untreated Childhood Myeloid Neoplasm
Keywords: Pediatrics; leukemia; invasive fungal infection
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Mycoses; Neutropenia; Leukemia; Invasive Fungal Infections | interventions — Caspofungin; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (caspofungin acetate) (Experimental): Patients receive caspofungin acetate IV over one hour QD beginning within 24-72 hours following the last dose of chemotherapy for each course. and continuing until ANC > 100-500/uL following the nadir or the next chemotherapy course begins.
  Interventions: Drug: Caspofungin Acetate; Other: Laboratory Biomarker Analysis
- Arm II (fluconazole) (Active Comparator): Patients receive fluconazole IV over 1-2 hours or PO QD beginning within 24-72 hours following the last dose of chemotherapy for each course.
  Interventions: Drug: Fluconazole; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Caspofungin Acetate — Given IV
  Other Names: Cancidas
  Arms: Arm I (caspofungin acetate)
Drug: Fluconazole — Given IV or PO
  Other Names: Diflucan
  Arms: Arm II (fluconazole)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase III trial compares the effectiveness of caspofungin to fluconazole in preventing invasive fungal infections in patients receiving chemotherapy for acute myeloid leukemia (AML). Antifungal prophylaxis is considered standard of care in children and adults with prolonged neutropenia after chemotherapy for AML however the ideal antifungal agent for prophylaxis in children is not known. Caspofungin has activity against yeast and some molds while fluconazole coverage is limited to just yeasts. Adult randomized trials suggest that agents with activity against yeasts and molds are more effective than those with just activity against yeasts. There are limited data to answer this comparative question in children. This study will establish much needed pediatric data to guide clinical decision making on optimal antifungal prophylaxis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if prophylaxis with caspofungin administered during periods of neutropenia following chemotherapy for acute myeloid leukemia (AML) is associated with a lower incidence of proven or probable invasive fungal infections (IFI) compared with fluconazole.

SECONDARY OBJECTIVES:

I. To determine if prophylaxis with caspofungin will result in a lower incidence of proven or probable cases of invasive aspergillosis (IA) compared with fluconazole. (Clinical) II. To determine if prophylaxis with caspofungin will result in improved survival compared to fluconazole. (Clinical) III. To determine if prophylaxis with caspofungin will result in less empiric antifungal therapy compared to fluconazole. (Clinical) IV. To determine the sensitivity, specificity, and positive and negative predictive value of biweekly galactomannan (GM) and beta-D glucan testing in diagnosing IFI. (Biological) V. To test the association between single nucleotide polymorphisms (SNPs) in genes involved in innate immunity and proven or probable IFI. (Biological) VI. To develop predictive models of IFI using SNP in genes involved in immunity and clinical covariates. (Biological)

OUTLINE: Patients are randomized to one of two treatment arms during their first chemotherapy course for AML.

ARM I: Patients receive caspofungin acetate intravenously (IV) over one hour once daily (QD) beginning within 24-72 hours following the last dose of chemotherapy for each course. and continuing until absolute neutrophil count (ANC) > 100-500/uL following the nadir or the next chemotherapy course begins.

ARM II: Patients receive fluconazole IV over 1-2 hours or orally (PO) QD beginning within 24-72 hours following the last dose of chemotherapy for each course.

Protocol prophylaxis was continued in both arms, until ANC increased to > 100-500/uL following the nadir or the next chemotherapy course began. Prophylaxis was given for all courses of planned AML chemotherapy or until the patient met one of the following off-protocol therapy criteria: development of proven or probable IFI according to institutional diagnosis, initiation of conditioning for hematopoietic cell transplantation, initiation of a new chemotherapy regimen for relapsed or refractory AML, refusal of further protocol therapy by patient, parent or guardian, or physician determines it is in the best interest of the patient.

Regardless of duration of prophylaxis, subjects in both arms are monitored for IFI until the earliest of the following criteria is met: two weeks after recovery of neutropenia following the last planned AML chemotherapy course, initiation of conditioning for hematopoietic cell transplantation, initiation of a new chemotherapy regimen for relapsed or refractory AML, withdrawal of consent for any further data submission, or death.

Patients were followed for overall survival up to two years from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following diagnoses and/or treatment plans:

  * Newly diagnosed de novo AML
  * First or subsequent relapse of AML
  * Secondary AML
  * Treatment with institutional standard AML therapy in those without AML (for example, myelodysplastic syndrome, bone marrow blasts > 5% or biphenotypia)
  * Note: Patients with a history of prolonged antifungal therapy (example, relapsed AML) are eligible
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR a serum creatinine based on age/gender as follows:

  * =< 0.4 mg/dL (age 1 month to < 6 months)
  * =< 0.5 mg/dL (age 6 months to < 1 year)
  * =< 0.6 mg/dL (age 1 to < 2 years)
  * =< 0.8 mg/dL (age 2 to < 6 years)
  * =< 1 mg/dL (age 6 to < 10 years)
  * =< 1.2 mg/dL (age 10 to < 13 years)
  * =< 1.4 mg/dL (females age >= 13 years)
  * =< 1.5 mg/dL (males age 13 to < 16 years)
  * =< 1.7 mg/dL (males age >= 16 years)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age AND Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x ULN for age
* All patients and/or their parents or legal guardians must sign a written informed consent

Exclusion Criteria:

* Patients with the following diagnoses are not eligible:

  * Acute promyelocytic leukemia (APL)
  * Down syndrome
  * Juvenile myelomonocytic leukemia (JMML)
* Patients with a documented history of invasive fungal infection (IFI) within the previous 30 days are not eligible
* Patients with a history of echinocandin or fluconazole hypersensitivity are not eligible
* Patients receiving treatment for an IFI are not eligible
* Female patients of childbearing age must have a negative pregnancy test
* Patients must agree to use an effective birth control method
* Lactating patients must agree not to nurse a child while on this trial

Ages: 3 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 517 (Actual)
Dates: Start 2011-04-04 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theoklis E Zaoutis, Principal Investigator — Children's Oncology Group
Locations (179):
- United States (166):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health Richland, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Fisher BT, Zaoutis T, Dvorak CC, Nieder M, Zerr D, Wingard JR, Callahan C, Villaluna D, Chen L, Dang H, Esbenshade AJ, Alexander S, Wiley JM, Sung L. Effect of Caspofungin vs Fluconazole Prophylaxis on Invasive Fungal Disease Among Children and Young Adults With Acute Myeloid Leukemia: A Randomized Clinical Trial. JAMA. 2019 Nov 5;322(17):1673-1681. doi: 10.1001/jama.2019.15702. PMID 31688884
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole)
Started | 257 | 260
Completed | 117 | 115
Not Completed | 140 | 145
Not completed — Death | 3 | 6
Not completed — Physician Decision | 26 | 29
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Institutional diagnosis of IFD | 21 | 36
Not completed — Begin conditioning for HSCT | 42 | 44
Not completed — Refractory or relapsed AML | 38 | 23
Not completed — Ineligible | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole) | Total
Number analyzed (Participants) | 257 | 260 | 517
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 235 | 242 | 477
  Between 18 and 65 years | 22 | 18 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: Years] | 9.2 (6.5) | 8.8 (6.0) | 9.0 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 114 | 228
  Male | 143 | 146 | 289
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 52 | 93
  Not Hispanic or Latino | 206 | 203 | 409
  Unknown or Not Reported | 10 | 5 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 19 | 19 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 29 | 32 | 61
  White | 181 | 179 | 360
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 27 | 26 | 53
Region of Enrollment [Number; unit: participants]
  United States | 234 | 227 | 461
  Canada | 22 | 33 | 55
  United Arab Emirates | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Proven or Probable Invasive Fungal Infections (IFI)
Description: Proven or probable IFI is defined according to criteria developed by the European Organization for Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG).
Time Frame: Up to 5 months since enrollment
Population: Evaluable patients (ineligible and inevaluable due to having IFI before IFI monitoring period were excluded)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole)
Number analyzed (Participants) | 253 | 255
Percentage of participants | 3.1 [1.3 to 7.0] | 7.2 [4.4 to 11.8]

2. Secondary Outcome: Percentage of Participants With Proven or Probable Invasive Aspergillosis (IA)
Description: Proven or probable invasive aspergillosis (IA) is defined according to the criteria developed by the EORTC/MSG. Kaplan Meier approach will used to estimate the incidence.
Time Frame: Up to 5 months since enrollment
Population: Evaluable patients (ineligible and inevaluable due to having IFI before IFI monitoring period were excluded)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole)
Number analyzed (Participants) | 253 | 255
Percentage of participants | 0.5 [0.1 to 3.5] | 3.1 [1.4 to 6.9]

3. Secondary Outcome: Overall Survival
Description: Kaplan Meier method will be used to estimate overall survival. Time to event is from enrollment to date of death (by any cause). Participants are censored at last contact or 2 years anniversary of enrollment into this study, whichever occurred first.
Time Frame: Up to 2 years post enrollment
Population: Evaluable patients (ineligible and inevaluable due to having IFI before IFI monitoring period were excluded)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole)
Number analyzed (Participants) | 253 | 255
Percentage of participants | 68.8 [62.3 to 74.4] | 70.8 [64.6 to 76.1]

4. Secondary Outcome: Percentage of Participants That Need Empiric Antifungal Therapy
Description: The percentage of participants requiring empiric antifungal therapy will be determined based on the presence of prolonged fever and neutropenia during each neutropenia course.
Time Frame: Up to 5 months since enrollment
Population: Evaluable patients (ineligible and inevaluable due to having IFI before IFI monitoring period were excluded)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole)
Number analyzed (Participants) | 253 | 255
Percentage of participants | 71.9 [65.1 to 78.4] | 69.5 [63.1 to 75.7]

5. Other Pre Specified Outcome: Sensitivity of Galactomannan and Beta-D Glucan Assays for the Diagnosis of Proven or Probable IFI
Description: Sensitivity for the diagnosis of proven or probable IFI will be determined for the fungal biomarkers galactomannan and beta-D glucan assays. Sensitivity will be estimated for the combination of the two fungal biomarkers.
Time Frame: Up to 5 months since enrollment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Specificity of Galactomannan and Beta-D Glucan Assays for the Diagnosis of Proven or Probable IFI
Description: Specificity of galactomannan and beta-D glucan assays for the diagnosis of proven or probable IFI. Specificity will be estimated for the two fungal biomarkers together.
Time Frame: Up to 5 months since enrollment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Positive Predictive Value of Galactomannan and Beta-D Glucan Assays for the Diagnosis of Proven or Probable IFI
Description: Positive predictive value of galactomannan and beta-D glucan assays for the diagnosis of proven or probable IFI. Positive predictive value will be estimated for the two fungal biomarkers together.
Time Frame: Up to 5 months since enrollment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Negative Predictive Value of Galactomannan and Beta-D Glucan Assays for the Diagnosis of Proven or Probable IFI
Description: Negative predictive value of galactomannan and beta-D glucan assays for the diagnosis of proven or probable IFI. Negative predictive value will be estimated for the two fungal biomarkers together.
Time Frame: Up to 5 months since enrollment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Genotyping Assays for Single Nucleotide Polymorphism Analysis
Description: Descriptive statistics will be used to summarize the prevalence of single nucleotide polymorphisms.
Time Frame: Up to 2 years post enrollment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 12 months of receiving protocol treatment
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Arm I (Caspofungin Acetate) | Arm II (Fluconazole)
All-Cause Mortality (participants affected / at risk) | 76/253 | 82/255
Serious Adverse Events (participants affected / at risk) | 11/253 | 9/255
Other Adverse Events (participants affected / at risk) | 62/253 | 72/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Caspofungin Acetate) (N=253) | Arm II (Fluconazole) (N=255)
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death NOS (General disorders) | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Edema cerebral (Nervous system disorders) | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Heart failure (Cardiac disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Investigations - Other, specify (Investigations) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0
Lung infection (Infections and infestations) | 1 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0
Multi-organ failure (General disorders) | 2 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural infection (Infections and infestations) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sepsis (Infections and infestations) | 2 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Caspofungin Acetate) (N=253) | Arm II (Fluconazole) (N=255)
Acute kidney injury (Renal and urinary disorders) | 0 | 3
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Alanine aminotransferase increased (Investigations) | 3 | 9
Allergic reaction (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 7
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 3
Cardiac arrest (Cardiac disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ejection fraction decreased (Investigations) | 1 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
Encephalitis infection (Infections and infestations) | 1 | 0
Encephalomyelitis infection (Infections and infestations) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 2
Fever (General disorders) | 4 | 1
GGT increased (Investigations) | 1 | 2
Heart failure (Cardiac disorders) | 2 | 4
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 20 | 11
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 3
Hypotension (Vascular disorders) | 12 | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 8 | 9
Investigations - Other, specify (Investigations) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 3
Lipase increased (Investigations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 2
Lymphocyte count decreased (Investigations) | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 3
Neutrophil count decreased (Investigations) | 4 | 1
Peritoneal infection (Infections and infestations) | 0 | 1
Platelet count decreased (Investigations) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Salivary gland infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 20 | 43
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Typhlitis (Gastrointestinal disorders) | 3 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
White blood cell decreased (Investigations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT01307579/Prot_SAP_000.pdf